CLINICAL TRIAL: NCT05710432
Title: Muscle Recruitment During Neck Flexion and Inspiratory Muscle Training in Difficult and Prolonged Weaning Patients: a Physiological Study - The FLEX Study
Brief Title: Muscle Recruitment During Neck Flexion and Inspiratory Muscle Training
Acronym: FLEX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 22-185
Record Dates: First submitted 2022-12-19; First posted 2023-02-02 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Mechanical Ventilator Weaning; Respiratory Muscle Training
Keywords: Mechanical Ventilation; Inspiratory Muscle Training; Neck Flexion; Mechanical Ventilator Weaning

STUDY DESIGN:
Intervention Model Description: As soon as patients can be disconnected from the ventilator and able to perform IMT, the order of the two training techniques (Quasi-isometric neck flexion exercise and inspiratory muscle training) will be randomized (using sealed opaque envelopes).
Who Masked: Investigator
Masking Description: The two training techniques will be randomized using sealed opaque envelopes.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quasi-Isometric Neck Flexion (Experimental): On minimal mechanical ventilation support (unassisted/assisted spontaneous breathing) via tracheostomy.
  Quasi-Isometric Neck Flexion will be performed during mechanical ventilation. Patients will be asked to minimally lift their head from the pillow generating a quasi-isometric neck contraction. 30% will be the target intensity level for neck flexion. The patient will perform 2 sets of 6-10 quasi-isometric neck flexions.
  Interventions: Other: Quasi-Isometric Neck Flexion; Other: Inspiratory Muscle Training
- Inspiratory Muscle Training (Experimental): Perform 2 sets of 6-10 breaths through a POWERbreathe device, which applies a variable resistance provided by an electronically controlled valve (variable flow resistive load). The training device will be set at 30% of the highest value of three MIP maneuvers. A two-minute rest period with MV support will be provided between each set.
  Interventions: Other: Quasi-Isometric Neck Flexion; Other: Inspiratory Muscle Training

INTERVENTIONS:
Other: Quasi-Isometric Neck Flexion — Patients will be asked to minimally lift their head from the pillow generating a quasi-isometric neck contraction (2 sets of 6-10 flexions).
Other: Inspiratory Muscle Training — Patients will be asked to complete 2 sets of 6-10 breaths through a POWERbreathe device, which applies a variable resistance provided by an electronically controlled valve (variable flow resistive load).
  During each IMT and neck flexion maneuver ultrasound measurements will be performed (measurements of the diaphragm, sternocleidomastoid, parasternal intercostal, internal oblique [IO], external oblique [EO], transversus abdominis [TrA] and rectus abdominis [RA] will be taken) and, during the entire period, sEMG monitoring of the target muscles (diaphragm, sternocleidomastoid, parasternal intercostal and EO) will be continued.

SUMMARY:
Respiratory muscle dysfunction is highly prevalent in patients with prolonged weaning from mechanical ventilation and is strongly associated with weaning failure. Efforts to strengthen the respiratory muscles, aimed at reversing or minimizing the impact of respiratory muscle weakness on clinical outcomes, have generally focused on the diaphragm with specific inspiratory muscle training (IMT) exercises. However, the effectiveness of these exercises and impact on clinical outcomes are not current practice in the majority of ICUs, as they are hardly feasible in ICU patients who often cannot be disconnected from the ventilator and cannot fully cooperate.

Promising results have been published concerning non-respiratory training techniques, which can also target the accessory muscles, particularly important in the presence of increased load to the respiratory system, as in the case of the weaning phase. These non-respiratory training techniques would have the advantage of not entailing disconnection of the patient from the ventilator. In particular, in healthy subjects, a quasi-isometric neck contraction, called neck flexion, appeared to generate greater or comparable recruitment of some principal and accessory muscles of respiration, when compared to conventional IMT. However, this has not been studied in patients requiring prolonged mechanical ventilation, for whom IMT with threshold loading devices remains the primary recommended rehabilitation strategy.

Therefore, the primary aim of the investigators is to assess the feasibility, tolerability, and safety of neck flexion and to compare them with IMT technique in patients with difficult and prolonged weaning from mechanical ventilation. Secondary aims are: i) to characterize which respiratory muscles are recruited and their level of activation at different levels of ventilatory assistance and ii) to assess which respiratory muscles are recruited and their level of activation during the two techniques and to compare these findings.

The hypothesis of the investigators is that neck flexion will be feasible (more than conventional IMT), well tolerated, and safe in patients with difficult and prolonged weaning. The investigators also hypothesize that, reducing the level of assistance and during unassisted breathing, a progressively increasing activation of the diaphragm, neck and trunk respiratory muscles, reflecting increased ventilatory load, will be fund. Finally, the hypothesis of the investigators is that the level of muscle activation/recruitment during neck flexion will be comparable or even greater to that occurring during IMT, as found in healthy subjects.

Finding a new and highly feasible rehabilitative technique, able to recruit and train the respiratory muscles (including accessory muscles), will have the potential to promote patients' weaning and improve all related clinical outcomes, and therefore to dramatically shift the paradigm about the role of rehabilitation in ICU.

DETAILED DESCRIPTION:
The investigators will conduct a prospective longitudinal pilot study in patients receiving mechanical ventilation via endotracheal tube or tracheostomy.

The investigators will perform a set of baseline measurements (as early as possible after the patient reaches the ability to spontaneously trigger the ventilator).These measurements include: I) ultrasound measurements (thickness and thickening fraction) of the diaphragm, parasternal intercostals, sternocleidomastoid and of the abdominal muscles; II) surface electromyography (sEMG) of the diaphragm, sternocleidomastoid, scalene, and of the abdominal muscles. Ultrasound and sEMG measurements will be performed during the current level of ventilation (decided by the clinical team), during minimal level of ventilatory support and/or during unassisted breathing; III) maximal inspiratory pressure (MIP); IV) maximal voluntary contraction (MVC) of neck flexion.

As soon as patients can be disconnected from the ventilator I) IMT maneuvers and II) neck flexion maneuvers, will be started and performed once a week (each time in a randomized order), until patients are successfully weaned or for a maximum of 4 weeks. The investigators will also perform: III) ultrasound measurements; IV) surface electromyography of the muscles above specified during each IMT and neck flexion maneuver; V) MIP and MVC; these latter measurements will be repeated weekly and inspiratory muscle training and neck flexion intensity level targeted accordingly.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving invasive MV via endotracheal tube who had failed a planned extubation or failed at least three spontaneous breathing trials (SBTs) or receiving MV via tracheostomy (who required tracheostomy because of difficult or prolonged weaning, failed extubation and/or prolonged ventilation) and able to spontaneously trigger the ventilator.
* Over or equal to 16 years of age
* Tolerating levels of pressure support of 10 cmH2O or lower (or equivalent support in NAVA or PAV+) for at least 15 minutes
* In stable clinical and hemodynamic conditions and adequate level of oxygenation (cardiac frequency ≤ 140 beats/minute, systolic blood pressure 90-160 mmHg, no or minimal vasopressors, PaO2/FiO2 over or equal to 150 mmHg)
* Able to understand and follow simple verbal instructions

Exclusion Criteria:

* Patients with a previously diagnosed severe neuromuscular disorder (such as amyotrophic lateral sclerosis, muscular dystrophy, multiple sclerosis, myasthenia gravis or spinal cord injury)
* Patients with chronic respiratory failure already ventilated before ICU admission
* Patients unable to collaborate or understand instructions

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-02-09 (Actual); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
Adherence to the training techniques | Baseline measurements assessed ≤ 72 hours from admission and once a week until successfully weaned or up to maximum of 4 weeks.
  Adherence to neck flexion and inspiratory muscle training techniques (minimum 70% completion), corresponding to the number of training sessions divided by the total number of potential sessions.
Incidence of Treatment-Emergent Adverse Events | Baseline measurements assessed ≤ 72 hours from admission and once a week until successfully weaned or up to maximum of 4 weeks.
  Neck flexion and IMT will be considered well tolerated if < 10% of patients refers dyspnea > 6 on the Borg scale (Borg scale minimum value is 0, which corresponds to no breathlessness at all; maximum value is 10, corresponding to the most severe breathlessness ever experienced or could imagine experiencing), or severe musculoskeletal soreness, during/after the training techniques.
  Neck flexion and IMT will be considered safe if < 5% of adverse events will be observed during/after the training techniques. Will be considered adverse events: desaturation over 4%, systolic blood pressure >180 mmHg or <90 mmHg or increased over or equal to 20%, cardiac arrhythmias, heart rate >140 beats/min or increased over or equal to 20%, respiratory rate >35 breaths/min or increased over or equal to 50%, cyanosis, diaphoresis, dizziness, facial signs of distress, evidence of increasing accessory muscle activity.

SECONDARY OUTCOMES:
Level of activation of the different respiratory muscles at different levels of ventilatory assistance through surface EMG | As early as possible after reaching the ability to spontaneously trigger the ventilator and tolerate a pressure support value of 10 cmH2O or below for at least 15 minutes until successfully weaned or a maximum of 4 weeks
  • To compare the level of activation during usual ventilatory setting vs minimal level of assistance/unassisted breathing paired t-test or Wilcoxon test will be performed.
Level of activation of the different respiratory muscles at different levels of ventilatory assistance through ultrasound | As early as possible after reaching the ability to spontaneously trigger the ventilator and tolerate a pressure support value of 10 cmH2O or below for at least 15 minutes until successfully weaned or a maximum of 4 weeks
  • To compare the level of activation during usual ventilatory setting vs minimal level of assistance/unassisted breathing paired t-test or Wilcoxon test will be performed.
Level of activation of the different respiratory muscles during the two training techniques (quasi-isometric neck flexion and IMT) through surface EMG | As early as possible after reaching the ability to spontaneously trigger the ventilator and tolerate a pressure support value of 10 cmH2O or below for at least 15 minutes until successfully weaned or a maximum of 4 weeks
  • To compare the degree of activation during IMT and neck flexion paired t-test or Wilcoxon test will be performed.
Level of activation of the different respiratory muscles during the two training techniques (quasi-isometric neck flexion and IMT) through ultrasound | As early as possible after reaching the ability to spontaneously trigger the ventilator and tolerate a pressure support value of 10 cmH2O or below for at least 15 minutes until successfully weaned or a maximum of 4 weeks
  • To compare the degree of activation during IMT and neck flexion paired t-test or Wilcoxon test will be performed.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beduneau G, Pham T, Schortgen F, Piquilloud L, Zogheib E, Jonas M, Grelon F, Runge I, Nicolas Terzi, Grange S, Barberet G, Guitard PG, Frat JP, Constan A, Chretien JM, Mancebo J, Mercat A, Richard JM, Brochard L; WIND (Weaning according to a New Definition) Study Group and the REVA (Reseau Europeen de Recherche en Ventilation Artificielle) Network double dagger. Epidemiology of Weaning Outcome according to a New Definition. The WIND Study. Am J Respir Crit Care Med. 2017 Mar 15;195(6):772-783. doi: 10.1164/rccm.201602-0320OC. PMID 27626706
- [Background] Boles JM, Bion J, Connors A, Herridge M, Marsh B, Melot C, Pearl R, Silverman H, Stanchina M, Vieillard-Baron A, Welte T. Weaning from mechanical ventilation. Eur Respir J. 2007 May;29(5):1033-56. doi: 10.1183/09031936.00010206. PMID 17470624
- [Background] Funk GC, Anders S, Breyer MK, Burghuber OC, Edelmann G, Heindl W, Hinterholzer G, Kohansal R, Schuster R, Schwarzmaier-D'Assie A, Valentin A, Hartl S. Incidence and outcome of weaning from mechanical ventilation according to new categories. Eur Respir J. 2010 Jan;35(1):88-94. doi: 10.1183/09031936.00056909. Epub 2009 Jun 18. PMID 19541716
- [Background] Herridge MS, Chu LM, Matte A, Tomlinson G, Chan L, Thomas C, Friedrich JO, Mehta S, Lamontagne F, Levasseur M, Ferguson ND, Adhikari NK, Rudkowski JC, Meggison H, Skrobik Y, Flannery J, Bayley M, Batt J, Santos CD, Abbey SE, Tan A, Lo V, Mathur S, Parotto M, Morris D, Flockhart L, Fan E, Lee CM, Wilcox ME, Ayas N, Choong K, Fowler R, Scales DC, Sinuff T, Cuthbertson BH, Rose L, Robles P, Burns S, Cypel M, Singer L, Chaparro C, Chow CW, Keshavjee S, Brochard L, Hebert P, Slutsky AS, Marshall JC, Cook D, Cameron JI; RECOVER Program Investigators (Phase 1: towards RECOVER); Canadian Critical Care Trials Group. The RECOVER Program: Disability Risk Groups and 1-Year Outcome after 7 or More Days of Mechanical Ventilation. Am J Respir Crit Care Med. 2016 Oct 1;194(7):831-844. doi: 10.1164/rccm.201512-2343OC. PMID 26974173
- [Background] Unroe M, Kahn JM, Carson SS, Govert JA, Martinu T, Sathy SJ, Clay AS, Chia J, Gray A, Tulsky JA, Cox CE. One-year trajectories of care and resource utilization for recipients of prolonged mechanical ventilation: a cohort study. Ann Intern Med. 2010 Aug 3;153(3):167-75. doi: 10.7326/0003-4819-153-3-201008030-00007. PMID 20679561
- [Background] Damuth E, Mitchell JA, Bartock JL, Roberts BW, Trzeciak S. Long-term survival of critically ill patients treated with prolonged mechanical ventilation: a systematic review and meta-analysis. Lancet Respir Med. 2015 Jul;3(7):544-53. doi: 10.1016/S2213-2600(15)00150-2. Epub 2015 May 20. PMID 26003390
- [Background] Claxton AR, Wong DT, Chung F, Fehlings MG. Predictors of hospital mortality and mechanical ventilation in patients with cervical spinal cord injury. Can J Anaesth. 1998 Feb;45(2):144-9. doi: 10.1007/BF03013253. PMID 9512849
- [Background] Dres M, Dube BP, Mayaux J, Delemazure J, Reuter D, Brochard L, Similowski T, Demoule A. Coexistence and Impact of Limb Muscle and Diaphragm Weakness at Time of Liberation from Mechanical Ventilation in Medical Intensive Care Unit Patients. Am J Respir Crit Care Med. 2017 Jan 1;195(1):57-66. doi: 10.1164/rccm.201602-0367OC. PMID 27310484
- [Background] Kim WY, Suh HJ, Hong SB, Koh Y, Lim CM. Diaphragm dysfunction assessed by ultrasonography: influence on weaning from mechanical ventilation. Crit Care Med. 2011 Dec;39(12):2627-30. doi: 10.1097/CCM.0b013e3182266408. PMID 21705883
- [Background] Jung B, Moury PH, Mahul M, de Jong A, Galia F, Prades A, Albaladejo P, Chanques G, Molinari N, Jaber S. Diaphragmatic dysfunction in patients with ICU-acquired weakness and its impact on extubation failure. Intensive Care Med. 2016 May;42(5):853-861. doi: 10.1007/s00134-015-4125-2. Epub 2015 Nov 16. PMID 26572511
- [Background] Goligher EC, Dres M, Fan E, Rubenfeld GD, Scales DC, Herridge MS, Vorona S, Sklar MC, Rittayamai N, Lanys A, Murray A, Brace D, Urrea C, Reid WD, Tomlinson G, Slutsky AS, Kavanagh BP, Brochard LJ, Ferguson ND. Mechanical Ventilation-induced Diaphragm Atrophy Strongly Impacts Clinical Outcomes. Am J Respir Crit Care Med. 2018 Jan 15;197(2):204-213. doi: 10.1164/rccm.201703-0536OC. PMID 28930478
- [Background] Goligher EC, Fan E, Herridge MS, Murray A, Vorona S, Brace D, Rittayamai N, Lanys A, Tomlinson G, Singh JM, Bolz SS, Rubenfeld GD, Kavanagh BP, Brochard LJ, Ferguson ND. Evolution of Diaphragm Thickness during Mechanical Ventilation. Impact of Inspiratory Effort. Am J Respir Crit Care Med. 2015 Nov 1;192(9):1080-8. doi: 10.1164/rccm.201503-0620OC. PMID 26167730
- [Background] Dres M, Goligher EC, Heunks LMA, Brochard LJ. Critical illness-associated diaphragm weakness. Intensive Care Med. 2017 Oct;43(10):1441-1452. doi: 10.1007/s00134-017-4928-4. Epub 2017 Sep 15. PMID 28917004
- [Background] Vorona S, Sabatini U, Al-Maqbali S, Bertoni M, Dres M, Bissett B, Van Haren F, Martin AD, Urrea C, Brace D, Parotto M, Herridge MS, Adhikari NKJ, Fan E, Melo LT, Reid WD, Brochard LJ, Ferguson ND, Goligher EC. Inspiratory Muscle Rehabilitation in Critically Ill Adults. A Systematic Review and Meta-Analysis. Ann Am Thorac Soc. 2018 Jun;15(6):735-744. doi: 10.1513/AnnalsATS.201712-961OC. PMID 29584447
- [Background] Elkins M, Dentice R. Inspiratory muscle training facilitates weaning from mechanical ventilation among patients in the intensive care unit: a systematic review. J Physiother. 2015 Jul;61(3):125-34. doi: 10.1016/j.jphys.2015.05.016. Epub 2015 Jun 16. PMID 26092389
- [Background] Martin AD, Smith BK, Davenport PD, Harman E, Gonzalez-Rothi RJ, Baz M, Layon AJ, Banner MJ, Caruso LJ, Deoghare H, Huang TT, Gabrielli A. Inspiratory muscle strength training improves weaning outcome in failure to wean patients: a randomized trial. Crit Care. 2011;15(2):R84. doi: 10.1186/cc10081. Epub 2011 Mar 7. PMID 21385346
- [Background] Gosselink R, De Vos J, van den Heuvel SP, Segers J, Decramer M, Kwakkel G. Impact of inspiratory muscle training in patients with COPD: what is the evidence? Eur Respir J. 2011 Feb;37(2):416-25. doi: 10.1183/09031936.00031810. PMID 21282809
- [Background] Hoffman M, Van Hollebeke M, Clerckx B, Muller J, Louvaris Z, Gosselink R, Hermans G, Langer D. Can inspiratory muscle training improve weaning outcomes in difficult to wean patients? A protocol for a randomised controlled trial (IMweanT study). BMJ Open. 2018 Jun 30;8(6):e021091. doi: 10.1136/bmjopen-2017-021091. PMID 29961023
- [Background] De Troyer A, Estenne M. Coordination between rib cage muscles and diaphragm during quiet breathing in humans. J Appl Physiol Respir Environ Exerc Physiol. 1984 Sep;57(3):899-906. doi: 10.1152/jappl.1984.57.3.899. PMID 6238017
- [Background] De Troyer A, Boriek AM. Mechanics of the respiratory muscles. Compr Physiol. 2011 Jul;1(3):1273-300. doi: 10.1002/cphy.c100009. PMID 23733642
- [Background] Shi ZH, Jonkman A, de Vries H, Jansen D, Ottenheijm C, Girbes A, Spoelstra-de Man A, Zhou JX, Brochard L, Heunks L. Expiratory muscle dysfunction in critically ill patients: towards improved understanding. Intensive Care Med. 2019 Aug;45(8):1061-1071. doi: 10.1007/s00134-019-05664-4. Epub 2019 Jun 24. PMID 31236639
- [Background] Laghi F, Shaikh HS, Morales D, Sinderby C, Jubran A, Tobin MJ. Diaphragmatic neuromechanical coupling and mechanisms of hypercapnia during inspiratory loading. Respir Physiol Neurobiol. 2014 Jul 1;198:32-41. doi: 10.1016/j.resp.2014.03.004. Epub 2014 Apr 16. PMID 24747754
- [Background] Ishida H, Suehiro T, Kurozumi C, Ono K, Watanabe S. Correlation Between Abdominal Muscle Thickness and Maximal Expiratory Pressure. J Ultrasound Med. 2015 Nov;34(11):2001-5. doi: 10.7863/ultra.14.12006. Epub 2015 Sep 22. PMID 26396169
- [Background] Dres M, Dube BP, Goligher E, Vorona S, Demiri S, Morawiec E, Mayaux J, Brochard L, Similowski T, Demoule A. Usefulness of Parasternal Intercostal Muscle Ultrasound during Weaning from Mechanical Ventilation. Anesthesiology. 2020 May;132(5):1114-1125. doi: 10.1097/ALN.0000000000003191. PMID 32084029
- [Background] Shi ZH, de Vries H, de Grooth HJ, Jonkman AH, Zhang Y, Haaksma M, van de Ven PM, de Man AAME, Girbes A, Tuinman PR, Zhou JX, Ottenheijm C, Heunks L. Changes in Respiratory Muscle Thickness during Mechanical Ventilation: Focus on Expiratory Muscles. Anesthesiology. 2021 May 1;134(5):748-759. doi: 10.1097/ALN.0000000000003736. PMID 33711154
- [Background] Vivier E, Roussey A, Doroszewski F, Rosselli S, Pommier C, Carteaux G, Mekontso Dessap A. Atrophy of Diaphragm and Pectoral Muscles in Critically Ill Patients. Anesthesiology. 2019 Sep;131(3):569-579. doi: 10.1097/ALN.0000000000002737. PMID 31094757
- [Background] Schreiber AF, Bertoni M, Coiffard B, Fard S, Wong J, Reid WD, Brochard LJ, Piva S, Goligher EC. Abdominal Muscle Use During Spontaneous Breathing and Cough in Patients Who Are Mechanically Ventilated: A Bi-center Ultrasound Study. Chest. 2021 Oct;160(4):1316-1325. doi: 10.1016/j.chest.2021.05.053. Epub 2021 Jun 6. PMID 34090872
- [Background] Enriquez D, Gomez Traverso R, Brizuela S, Szyld E. [Mistakes in drug prescription during simulated pediatric resuscitations and other urgency procedures]. Arch Argent Pediatr. 2017 Jun 1;115(3):294-299. doi: 10.5546/aap.2017.294. Spanish. PMID 28504508
- [Background] DePalo VA, Parker AL, Al-Bilbeisi F, McCool FD. Respiratory muscle strength training with nonrespiratory maneuvers. J Appl Physiol (1985). 2004 Feb;96(2):731-4. doi: 10.1152/japplphysiol.00511.2003. Epub 2003 Sep 26. PMID 14514702
- [Background] Derbakova A, Khuu S, Ho K, Lewis C, Ma T, Melo LT, Zabjek KF, Goligher EC, Brochard L, Fregonezi G, Reid WD. Neck and Inspiratory Muscle Recruitment during Inspiratory Loading and Neck Flexion. Med Sci Sports Exerc. 2020 Jul;52(7):1610-1616. doi: 10.1249/MSS.0000000000002271. PMID 31977643
- [Background] Goligher EC, Laghi F, Detsky ME, Farias P, Murray A, Brace D, Brochard LJ, Bolz SS, Rubenfeld GD, Kavanagh BP, Ferguson ND. Measuring diaphragm thickness with ultrasound in mechanically ventilated patients: feasibility, reproducibility and validity. Intensive Care Med. 2015 Apr;41(4):642-9. doi: 10.1007/s00134-015-3687-3. Epub 2015 Feb 19. PMID 25693448
- [Background] Matamis D, Soilemezi E, Tsagourias M, Akoumianaki E, Dimassi S, Boroli F, Richard JC, Brochard L. Sonographic evaluation of the diaphragm in critically ill patients. Technique and clinical applications. Intensive Care Med. 2013 May;39(5):801-10. doi: 10.1007/s00134-013-2823-1. Epub 2013 Jan 24. PMID 23344830
- [Background] Formenti P, Umbrello M, Dres M, Chiumello D. Ultrasonographic assessment of parasternal intercostal muscles during mechanical ventilation. Ann Intensive Care. 2020 Sep 7;10(1):120. doi: 10.1186/s13613-020-00735-y. PMID 32894372
- [Background] Hong BY, Ko YJ, Kim JS, Ok EJ, Hwang Y, Kim HW. Sternocleidomastoid ultrasonography data for muscular torticollis in infants. Muscle Nerve. 2013 Jul;48(1):100-4. doi: 10.1002/mus.23712. Epub 2013 Apr 21. PMID 23605885
- [Background] Kubas C, Chen YW, Echeverri S, McCann SL, Denhoed MJ, Walker CJ, Kennedy CN, Reid WD. Reliability and Validity of Cervical Range of Motion and Muscle Strength Testing. J Strength Cond Res. 2017 Apr;31(4):1087-1096. doi: 10.1519/JSC.0000000000001578. PMID 27467513
- [Background] Marini JJ, Smith TC, Lamb V. Estimation of Inspiratory Muscle Strength in Mechanically Ventilated Patients: The Measurement of Maxima Inspiratory Pressure. J Crit Care. 1986;1(1):32-8.
- [Background] de Almeida LB, Trevizan PF, Laterza MC, Hallack Neto AE, Perrone ACASJ, Martinez DG. Safety and feasibility of inspiratory muscle training for hospitalized patients undergoing hematopoietic stem cell transplantation: a randomized controlled study. Support Care Cancer. 2020 Aug;28(8):3627-3635. doi: 10.1007/s00520-019-05209-x. Epub 2019 Dec 5. PMID 31807987
- [Background] Fioritto AP, Oliveira CC, Albuquerque VS, Almeida LB, Granger CL, Denehy L, Malaguti C. Individualized in-hospital exercise training program for people undergoing hematopoietic stem cell transplantation: a feasibility study. Disabil Rehabil. 2021 Feb;43(3):386-392. doi: 10.1080/09638288.2019.1626493. Epub 2019 Jun 11. PMID 31184516